CLINICAL TRIAL: NCT04133662
Title: Sleep and Pain in Childhood Arthritis: A Crossover Randomized Trial Comparing Adequate and Restricted Sleep Duration, and Its Impact on Pain in Adolescents With Arthritis
Brief Title: Sleep & Pain in Juvenile Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Brian Feldman, Division Head, Division of Rheumatology, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1000061386
Record Dates: First submitted 2019-10-08; First posted 2019-10-21 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Arthritis, Juvenile
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Restricted sleep condition first, longer sleep condition second
  Interventions: Behavioral: Sleep Manipulation Protocol
- Group 2 (Experimental): Longer sleep condition first, restricted sleep condition second
  Interventions: Behavioral: Sleep Manipulation Protocol

INTERVENTIONS:
Behavioral: Sleep Manipulation Protocol — A structured sleep duration intervention will be taught to patients

SUMMARY:
Childhood arthritis is an important cause of pain for affected children and youth (adolescents). Many youth with arthritis also have trouble sleeping. They often struggle to sleep through the night, wake up earlier, and are sleepier during the day compared to healthy children. Our research group, among others, has shown a strong link between sleep and pain. The main purpose of this study is to assess the impact of changing sleeping patterns on pain, and disease activity, in teenagers with arthritis. We think that better sleep will directly lead to better health.

ELIGIBILITY:
Inclusion Criteria:

* patient in the rheumatology clinic at SickKids
* all subtypes of JIA, as per the ILAR criteria
* a baseline pain score of ≥ 1 on a visual analogue scale
* age from 12-18 years old
* capable of providing informed consent form themselves, as judged by the clinical team

Exclusion Criteria:

* a known sleep disorder (e.g., obstructive sleep apnea, etc.)
* a high probability of having obstructive sleep apnea as determined by the Pediatric Sleep Questionnaire
* currently taking medication with the intent to impact sleep (e.g., zolpidem, benzodiazepines, etc.)
* taking corticosteroids (which may adversely affect sleep)
* obligations that require a bed time later than 10:00 pm or a wake time earlier than 5:30 am during the study period
* daily consumption of > 1 coffee or "energy drink" and/or > 3 caffeinated carbonated beverages
* do not speak/understand English with enough proficiency to complete all study related tasks, as judged by the clinical team

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
Change in Pain as measured on the PROMIS Pain Interference Scale | baseline, end of baseline week, end of experimental week 1, end of experimental week 2
  Change in Pain as measured on the PROMIS (Patient-Reported Outcomes Measurement Information System) Pain Interference Scale. Scores can range from 0-100 with 100 representing the best possible outcome

SECONDARY OUTCOMES:
Change in Pain as measured on the PROMIS Pain Behaviour Scale | baseline, end of baseline week, end of experimental week 1, end of experimental week 2
  Change in Pain as measured on the PROMIS (Patient-Reported Outcomes Measurement Information System) Pain Behaviour Scale. Scores can range from 0-100 with 100 representing the best possible outcome
Pain as measured using the iCanCope with Pain app | end of study (3 weeks)
  Pain as measured using the iCanCope with Pain app
Change in Disease Activity | baseline, end of baseline week, end of experimental week 1, end of experimental week 2
  measured using the clinical Juvenile Arthritis Disease Activity Score (JADAS). Scored on a scale from 0-27, with 0 representing the best possible outcome
Change in Functional Status | baseline, end of baseline week, end of experimental week 1, end of experimental week 2
  measured using the Childhood Health Assessment Questionnaire (CHAQ). Scored on a scale of 0-3, with 0 representing the best possible outcome.
Change in Health Related Quality of Life | baseline, end of baseline week, end of experimental week 1, end of experimental week 2
  measured using the Quality of My Life (QoML) questionnaire. This measure is comprised of 2 visual analog scales that measure overall quality of life and health related quality of life. Each scale ranges from 0-10 with 10 representing the best possible outcome.
Physical Activity | end of study (3 weeks)
  measured using a wrist-mounted accelerometer, we will measure the amount of time the subjects spend sedentary, mild, moderate to vigorous (MVPA), and vigorous (VPA) physical activity by looking at total metabolic equivalents (METs).
Change in Inattention and Sleepiness | baseline, end of baseline week, end of experimental week 1, end of experimental week 2
  measured using the Inattention and Sleepiness Behaviour Rating Scale, scored on a scale of 0-39 with 0 representing the best possible score. Each sub-section can also be scored individually, with sleepiness being scored on a scale of 0-15 and inattention being scored on a scale of 0-27, with 0 representing the best possible score in both cases (i.e. the least sleepiness and least inattention)

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clairman H, Dover S, Tomlinson G, Beebe D, Cameron B, Laxer RM, Levy D, Narang I, Paetkau S, Schneider R, Spiegel L, Stephens S, Stinson J, Tse S, Weiss S, Whitney K, Feldman BM. Lengthening sleep reduces pain in childhood arthritis: a crossover randomised controlled trial. RMD Open. 2023 Oct;9(4):e003352. doi: 10.1136/rmdopen-2023-003352. PMID 37914178